CLINICAL TRIAL: NCT01420094
Title: Comparative Onset of Action of a Fast Release Aspirin Tablet in a Dental Impaction Pain Model
Brief Title: Evaluate Onset of Action of a Fast Release Aspirin
Acronym: TAROT compare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15529; 2014-005270-11 (EudraCT Number)
Record Dates: First submitted 2011-07-27; First posted 2011-08-19 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Healthy Subjects
Keywords: Drugs, Investigational; Acetylsalicylic Acid; Aspirin; dental pain
MeSH Terms: conditions — Toothache | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicyclic acid (Fast release Aspirin, BAY1019036)
- Arm 2 (Active Comparator)
  Interventions: Drug: Acetaminophen (Tylenol extra strength)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicyclic acid (Fast release Aspirin, BAY1019036) — Single oral dose of fast release aspirin tablet 1000 mg (2 x 500 mg) and 2 placebo-matching acetaminophen caplets with a full glass of water (240 milliliter [mL]) between 1-4 hours post dental surgery.
  Arms: Arm 1
Drug: Acetaminophen (Tylenol extra strength) — Single oral dose of acetaminophen (Tylenol extra strength) caplet 1000 mg (2 x 500 mg) and 2 placebo matching aspirin tablets with a full glass of water (240 mL) between 1-4 hours post dental surgery.
  Arms: Arm 2
Drug: Placebo — Single oral dose of placebo (2 placebo aspirin tablets and 2 placebo acetaminophen caplets) with a full glass of water (240 mL) between 1-4 hours post dental surgery.
  Arms: Arm 3

SUMMARY:
To compare the safety and efficacy (onset, duration of relief and overall efficacy) of a single dose of a fast release formulation of aspirin 1000 mg compared to acetaminophen 1000 mg and placebo for relief of pain following extraction of impacted third molars.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers between 16 to 45 years of age
* Scheduled to undergo surgical removal of either two partial bony impactions or one full bony alone or in combination with a partial bony impaction, soft tissue impaction or erupted third molar. Maxillary third molars may be removed regardless of impaction level
* Use of only short-acting local anesthetic (e.g., mepivacaine or lidocaine) preoperatively, with or without vasoconstrictor and nitrous oxide
* No use of any analgesics, nonsteroidal anti-inflammatory drug (NSAIDs), aspirin, any other pain reliever over the counter (OTC ) or prescription, or herbal supplements within 5 days of surgery. Oral contraceptives, prophylactic antibiotics, pre-anesthetic medication, anesthesia during the procedure, or other routine medications to treat benign conditions that would not confound the evaluation of the investigational would be acceptable
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, NuvaRing, Depo-Provera, or double-barrier and have a negative pregnancy test at Screening and prior to surgery. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial, (subjects < 18 years of age must sign a written assent and have parental or guardian consent)

Exclusion Criteria:

* History of hypersensitivity to aspirin, salicylates, other nonsteroidal anti-inflammatory drug (NSAIDs), acetaminophen, opioid analgesics, and similar pharmacological agents or components of the investigational products, including the placebo
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than 50 percent obstruction (polyposis nasi, marked septal deviation) that can interfere with the conduct of the study in the judgment of the Investigator
* Current or past history of bleeding disorder(s)
* History of gastrointestinal bleeding or perforation, related to previous nonsteroidal anti-inflammatory drug (NSAID) therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Acute illness or local infection prior to surgery that can interfere with the conduct of the study in the judgment of the Investigator
* Females who are pregnant or lactating
* Positive alcohol breathalyzer test and/or positive urine drug or cotinine test prior to surgery

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 510 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2011-09-08 (Actual); Study Completion 2011-09-08 (Actual)

PRIMARY OUTCOMES:
Time to Meaningful Pain Relief (PR) | 0 to 6 hours

SECONDARY OUTCOMES:
Time to First Perceptible Pain Relief | 0 to 6 hours
Time to First Perceptible Pain Relief Confirmed | 0 to 6 hours
Pain Intensity at 5, 10, 15, 20, 25, 30, 35, 40, 50, and 60 minutes and at 1.5, 2, 3, 4, 5, and 6 hours After Dosing | 5, 10, 15, 20, 25, 30, 35, 40, and 50 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours post-dose
Pain Relief at 5, 10, 15, 20, 25, 30, 35, 40, 50, and 60 minutes and at 1.5, 2, 3, 4, 5, and 6 hours After Dosing | 5, 10, 15, 20, 25, 30, 35, 40, and 50 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours After Dosing
Pain Intensity Difference (PID) at 5, 10, 15, 20, 25, 30, 35, 40, 50, and 60 minutes and at 1.5, 2, 3, 4, 5, and 6 hours After Dosing | 5, 10, 15, 20, 25, 30, 35, 40, and 50 minutes and 1, 1.5, 2, 3, 4, 5, and 6 hours
Summed Pain Intensity Differences (SPID) from Hour 0 through Hour 2, Hour 4 and Hour 6 | 0 - 6 hours post-dose
Summed Total Pain Relief (TOTPAR) from Hour 0 through Hour 2, Hour 4 and Hour 6 | 0 to 6 hours post-dose
Time to First use of Rescue Medication | 0 to 6 hours
Cumulative Percentage of Subjects Taking Rescue Medication | 1, 2, 3, 4, 5, and 6 hours post-dose
Global Assessment of the Investigational Product as a Pain Reliever at 6 hours After Dosing or Immediately Before the First Intake of Rescue Medication | At 6 hours postdose or immediately before first use of rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Voelker M, Schachtel BP, Cooper SA, Gatoulis SC. Efficacy of disintegrating aspirin in two different models for acute mild-to-moderate pain: sore throat pain and dental pain. Inflammopharmacology. 2016 Feb;24(1):43-51. doi: 10.1007/s10787-015-0253-0. Epub 2015 Nov 24. PMID 26603742
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/